CLINICAL TRIAL: NCT01339195
Title: Post-stroke Cognitive Impairment and Dementia: Frequency and Anatomical Correlates With the French Version of the National Institute of Neurological Disorders and Stroke (NINDS)-Canadian Stroke Network Battery
Brief Title: Post-stroke Cognitive Impairment and Dementia
Acronym: GRECogVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOL10-PR-GODEFROY; 2010-A00657-32 (Other: CHU)
Record Dates: First submitted 2011-02-22; First posted 2011-04-20 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Cognitive Disorders; Behavioral Disorders
Keywords: Dementia; Alzheimer disease; stroke; cognitive impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Mental Disorders; Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral (Experimental): Behavioral: French adaptation of NINDS-Canadian Stroke Network battery
  Interventions: Behavioral: French adaptation of NINDS-Canadian Stroke Network battery

INTERVENTIONS:
Behavioral: French adaptation of NINDS-Canadian Stroke Network battery — * clinical: post-stroke neurological follow-up assessment
  * neuropsychological: comprising the NINDS-Canadian Stroke Network neuropsychological battery
  * MRI

SUMMARY:
Projections from epidemiological studies suggest that, among the Western adult population, one in three will present a cerebrovascular accident (stroke), severe cognitive disorders, or both. To better diagnose the Vascular Cognitive Impairment, new standards were developed by a North America working group which are under validation. It is essential to adapt these standard for French-speaking population, and especially to define cutoff scores of the cognitive battery to determine cognitive deficit.

The investigators propose a study coordinated by the University-Hospital of Amiens for french speaking centers. This study will investigate this battery with 906 controls to define the standards and 302 stroke affected patients to define the frequency and cognitive mechanisms. This step is essential for people to benefit from these new standards.

DETAILED DESCRIPTION:
* Context In western countries, one in three subjects will experience a stroke, dementia or both. Recent studies have shown the major role of vascular risk factors and stroke in cognitive disorders and dementia. Poststroke cognitive and behavioral disorders are characterized by the prominence of action slowing, executive function disorders and apathy. They are due to vascular lesions or to associated pathology, mainly Alzheimer's disease. In order to determine diagnosis criteria of Vascular Cognitive Impairment, it is necessary to develop a standardized assessment of post-stroke cognitive and behavioral disorders (Hachinski et al Stroke 2006; 37; 2220-2241). For this purpose, the NINDS (National Institute of Neurological Disorders and Stroke

  ) and the Canadian Stroke Network have jointly developed a specific standardized battery which is currently under validation. Its use in France requires first a normalization of some tests in French speaking healthy controls. This study is supported by the SFNV (Société Française NeuroVasculaire) and GRECO (Groupe de Réflexion sur les Evaluations Cognitives).
* Primary Objectives of the project: to determine the frequency of cognitive and behavioral disorders 6 months post-stroke assessed with this new NINDS-Canadian Stroke Network battery Primary endpoints: disorders on cognitive tests and on behavioral and depression questionnaires (defined by performance outside normal ranges determined in healthy controls);
* Population Patients consecutive French-speaking patients with an informant assessed 6 months post-stroke and free from mental retardation, psychosis, illiteracy, previously diagnosed dementia, comorbidity known to impair cognitive abilities, MRI contraindication or refusal to participate.

Controls from the general population not presenting any condition known to impair cognitive abilities stratified according to age and schooling levels

* Design Prospective multicenter study comparing performance of patients and controls Sample size: the frequencies of cognitive and behavioral disorders are considered as significantly different if the null hypothesis (lack of difference between groups at the 0.05 quantile) is rejected. Considering that each patient is matched with 3 controls, it will be necessary to evaluate 302 patients with the battery 6 months poststroke and 906 controls to detect a difference between groups of at least 5% with α risk =0.05 and power= 80%. In addition, the inclusion of 302 patients allows to determine the frequency of impaired patients with a confidence interval CI95% ≤12%.
* Feasibility: based on a previous similar study, 50 stroke patients (range 40-60) and 150 controls (range: 100-200) will be included per year in the University Hospital of Amiens. Thus 10 centers with similar inclusion rates will be able to include 302 patients and 906 controls within 6 years.
* Secondary objectives: (1) to determine the frequency of poststroke dementia; (2) to determine the frequency of cognitive disorders on screening tests; (3) to examine correlations between cerebral MRI and cognitive impairment; (4) to determine correlations between cognitive disorders and activities of daily living.

Secondary endpoints: (1) dementia (DSMIV and NINDS-AIREN criteria ;National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences ); (2) screening tests (MiniMental Status Examination, Montreal Cognitive Assessment);(3) MRI abnormalities (cerebral atrophy, white matter abnormalities, stroke type, stroke volume and location) using 3D T1-weighted (axial bicommissural plane), T2-weighted (coronal plan), FLAIR, gradient-echo, diffusion-weighted (with calculation of the apparent diffusion coefficient) performed at 6 months post-stroke at the same time than the cognitive assessment; (4) disability in activities of daily living (Rankin scale, Barthel index, Instrumental Activities of Daily Living).

ELIGIBILITY:
Inclusion criteria:

* Patients:management at the acute phase (duration < 30 days) of stroke visualized by imaging, age between 40 and 80 years, French-speaking, reliable informant, agreeing to participate in the study.
* Controls: derived from the general population and consenting to participate in the study.

Exclusion criteria:

* Patients: mental retardation, illiteracy, known dementia, schizophrenia or psychosis or history of psychiatric illness requiring a stay for > 2 days in a psychiatry unit, comorbidities affecting cognition, persistent disturbance of consciousness, contraindication to MRI.
* Controls: illiteracy, deficit on MMSE (Mini-Mental State Examination), visual, auditory or motor deficit, history of brain disease or psychiatric illness (schizophrenia or other psychosis) or ongoing psychiatric illness (depression or other) currently requiring treatment or requiring a stay > 2 days in psychiatry unit or anxiety requiring more than one medication at the present time, alcoholism, opiate or illicit drug use < 3 months, ongoing antidepressant or antiepileptic treatment, recent anxiolytic or hypnotic treatment, general anaesthesia < 3 months, history of heart surgery with cardiopulmonary bypass

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1635 (Actual)
Dates: Start 2010-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
determine the frequency of cognitive and behavioral disorders 6 months post-stroke assessed with this new NINDS-Canadian Stroke Network battery | 6 month
  deficit (as compared with control performance) on battery of tests assessing instrumental (oral naming, copy of complex figure)and executive fucntions (verbal fluency, Trail Making, reaction time tests), episodic memory for verbal and visual materials and behavioral changes

SECONDARY OUTCOMES:
determine the proportion of patients with dementia | 6 month
  composite index including memory and cognitive disorders and decline in every day life activities
determine the value of cognitive screening tests | 6 month
  performance on MiniMental State Examination and Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Godefroy, PhD-MD, Study Chair — CHU Amiens; Hilde Henon, MD, Principal Investigator — CHRU LILLE; Hervé Taillia, PhD-MD, Principal Investigator — HIA val de grace; Serge Timsit, PhD-MD, Principal Investigator — CHU Brest; Claudine Nedelec, MD, Principal Investigator — CH La Rochelle; catherine thomas, MD, Principal Investigator — CHU SAINT-ETIENNE; Maurice Giroud, PhD-MD, Principal Investigator — CHU Dijon
Locations (7):
- France (7):
  - CHRU Lille, Lille, Pas-de-calais
  - CHU Amiens, Amiens, Picardie
  - CHU Brest, Brest
  - CHU Dijon, Dijon
  - CH La Rochelle, La Rochelle
  - HIA Val de Grâce, Paris
  - CHU Saint Etienne, Saint-Etienne

REFERENCES:
- [Background] Godefroy O, Fickl A, Roussel M, Auribault C, Bugnicourt JM, Lamy C, Canaple S, Petitnicolas G. Is the Montreal Cognitive Assessment superior to the Mini-Mental State Examination to detect poststroke cognitive impairment? A study with neuropsychological evaluation. Stroke. 2011 Jun;42(6):1712-6. doi: 10.1161/STROKEAHA.110.606277. Epub 2011 Apr 7. PMID 21474808
- [Background] Godefroy O, Just A, Ghitu A, Leclercq C, Garcia PY, Lamy C, Canaple S, Bugnicourt JM. The Rankin scale with revised structured interview: effect on reliability, grading of disability and detection of dementia. Int J Stroke. 2012 Feb;7(2):183. doi: 10.1111/j.1747-4949.2011.00743.x. No abstract available. PMID 22264374
- [Result] Godefroy O; GRECOG-VASC study group; Leclercq C, Bugnicourt JM, Roussel M, Moroni C, Quaglino V, Beaunieux H, Taillia H, Nedelec-Ciceri C, Bonnin C, Thomas-Anterion C, Varvat J, Aboulafia-Brakha T, Assal F. Neuropsychological assessment and cerebral vascular disease: the new standards. Rev Neurol (Paris). 2013 Oct;169(10):779-85. doi: 10.1016/j.neurol.2013.07.009. Epub 2013 Aug 30. PMID 23999023
- [Result] Godefroy O, Leclercq C, Roussel M, Moroni C, Quaglino V, Beaunieux H, Tallia H, Nedelec-Ciceri C, Bonnin C, Thomas-Anterion C, Varvat J, Aboulafia-Brakha T, Assal F; GRECOG-VASC Neuropsychological Committee. French adaptation of the vascular cognitive impairment harmonization standards: the GRECOG-VASC study. Int J Stroke. 2012 Jun;7(4):362-3. doi: 10.1111/j.1747-4949.2012.00794.x. No abstract available. PMID 22583525
- [Result] Barbay M, Taillia H, Nedelec-Ciceri C, Bompaire F, Bonnin C, Varvat J, Grangette F, Diouf M, Wiener E, Mas JL, Roussel M, Godefroy O; GRECOG-VASC Study Group. Prevalence of Poststroke Neurocognitive Disorders Using National Institute of Neurological Disorders and Stroke-Canadian Stroke Network, VASCOG Criteria (Vascular Behavioral and Cognitive Disorders), and Optimized Criteria of Cognitive Deficit. Stroke. 2018 May;49(5):1141-1147. doi: 10.1161/STROKEAHA.117.018889. Epub 2018 Apr 11. PMID 29643258
- [Result] Godefroy O, Yaiche H, Taillia H, Bompaire F, Nedelec-Ciceri C, Bonnin C, Varvat J, Vincent-Grangette F, Diouf M, Mas JL, Canaple S, Lamy C, Arnoux A, Leclercq C, Tasseel-Ponche S, Roussel M, Barbay M; GRECogVASC Study Group. Who should undergo a comprehensive cognitive assessment after a stroke? A cognitive risk score. Neurology. 2018 Nov 20;91(21):e1979-e1987. doi: 10.1212/WNL.0000000000006544. Epub 2018 Oct 17. PMID 30333160